CLINICAL TRIAL: NCT00001752
Title: Vascular and Metabolic Effects of Hormone Therapy Combined With L-Arginine in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980158; 98-H-0158
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Hypercholesterolemia; Postmenopause
Keywords: Adhesion Molecules; Endothelial Function; Inflammation; Lipoproteins; Nitric Oxide; Hormone Therapy; Postmenopausal Women
MeSH Terms: conditions — Hypercholesterolemia; Inflammation | interventions — Arginine; Estrogens

INTERVENTIONS:
Drug: L-arginine
Drug: Estrogen

SUMMARY:
Estrogen therapy has been associated with reduced risk of coronary heart disease events in observational studies of postmenopausal women. Although favorable effects of estrogen on lipoprotein cholesterol levels probably account for much of this benefit, direct vascular effects (vasomotor, hemostatic, anti-inflammatory) regulated by nitric oxide (NO) may also be of importance. We have recently shown that vasodilator effects of estrogen in the coronary circulation are due to enhanced bioactivity of NO released from the endothelium. Estrogen has been shown to stimulate synthesis and activity of the enzyme NO synthase with enhanced NO synthesis in endothelial cells in culture. Because L-arginine is the natural substrate for the enzyme NO synthase, we propose that the combination of L-arginine and estrogen might have additive vasomotor, hemostatic and anti-inflammatory effects in hypercholesterolemic postmenopausal women.

DETAILED DESCRIPTION:
Estrogen therapy has been associated with reduced risk of coronary heart disease events in observational studies of postmenopausal women. Although favorable effects of estrogen on lipoprotein cholesterol levels probably account for much of this benefit, direct vascular effects (vasomotor, hemostatic, anti-inflammatory) regulated by nitric oxide (NO) may also be of importance. We have recently shown that vasodilator effects of estrogen in the coronary circulation are due to enhanced bioactivity of NO released from the endothelium. Estrogen has been shown to stimulate synthesis and activity of the enzyme NO synthase with enhanced NO synthesis in endothelial cells in culture. Because L-arginine is the natural substrate for the enzyme NO synthase, we propose that the combination of L-arginine and estrogen might have additive vasomotor, hemostatic and anti-inflammatory effects in hypercholesterolemic postmenopausal women.

ELIGIBILITY:
All volunteer subjects will be assessed for study participation, including a cardiovascular physical examination and resting electrocardiogram. Fasting blood will be taken for SMAC, CBC, thyroid battery, lipid levels, estradiol and FSH levels under screening protocol 94-H-0045. A urine pregnancy test will be performed in women with a uterus and cessation of menses less than 6 months. Aspirin and non-steroidal anti-inflammatory drugs and steroidal drugs (oral, ointment, drops or inhalation) will be stopped 10 days prior to starting the study and discontinued throughout the study.

Thirty hypercholesterolemic (LDL greater than 130 mg/dL) postmenopausal women who have not taken estrogenic hormone, antioxidant vitamins (A, C, E), or lipid-lowering therapy in the preceding 2 months will be selected to take part in this double-blind, cross-over study.

No subjects with plasma estradiol level greater than 50 pg/ml and FSH less than 50 pg/ml.

No subjects with blood pressure greater than 160/100 mm/Hg (off medication).

No subjects smoking cigarettes within 6 months.

No pregnant subjects.

No subjects with a history of deep venous thrombosis/pulmonary embolus.

No subjects with important chronic medical conditions (cancer, coronary artery disease, diabetes mellitus, COPD, renal disease) other than hypothyroidism if the subject is euthyroid on thyroid replacement.

No subjects who refuse to follow nitrate-restricted diet for 3 days prior to each study.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 1998-09; Study Completion 2000-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Guetta V, Quyyumi AA, Prasad A, Panza JA, Waclawiw M, Cannon RO 3rd. The role of nitric oxide in coronary vascular effects of estrogen in postmenopausal women. Circulation. 1997 Nov 4;96(9):2795-801. doi: 10.1161/01.cir.96.9.2795. PMID 9386140
- [Background] Hayashi T, Fukuto JM, Ignarro LJ, Chaudhuri G. Basal release of nitric oxide from aortic rings is greater in female rabbits than in male rabbits: implications for atherosclerosis. Proc Natl Acad Sci U S A. 1992 Dec 1;89(23):11259-63. doi: 10.1073/pnas.89.23.11259. PMID 1454805